CLINICAL TRIAL: NCT01350336
Title: Post-FDA Approval Clinical Trial Evaluating Bronchial Thermoplasty in Severe Persistent Asthma
Brief Title: Bronchial Thermoplasty in Severe Persistent Asthma
Acronym: PAS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-02
Record Dates: First submitted 2011-04-15; First posted 2011-05-09 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alair (Experimental): Alair system
  Interventions: Device: Alair System

INTERVENTIONS:
Device: Alair System — Treatment of airways with the Alair System

SUMMARY:
As Conditions of Approval of the PMA for the Alair System, the FDA requires Boston Scientific to generate data to assess the durability of the BT treatment effect as well as safety data in the intended use population in the United States.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single arm study designed to demonstrate durability of the treatment effect and to evaluate the short-term and longer-term safety profile of the Alair System in the United States in the intended use population (patients 18 years and older with severe persistent asthma).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is an adult between the ages of 18 to 65 years.
2. Subject is able to read, understand, and sign a written Informed Consent to participate in the study and able to comply with the study protocol.
3. Subject has asthma and is taking regular maintenance medication that includes:

   1. Inhaled corticosteroid (ICS) at a dosage greater than 1000μg beclomethasone per day or equivalent, AND long acting β2-agonist (LABA) at a dosage of ≥80μg per day Salmeterol or equivalent.
   2. Other asthma medications such as leukotriene modifiers, or anti-IgE, are acceptable (Subjects on Xolair® must have been on Xolair for greater than 1 year).
   3. Oral corticosteroids (OCS) at a dosage of up to, but not greater than 10mg per day are acceptable.*
4. Subject has a pre-bronchodilator FEV1 of greater than or equal to 60% of predicted.
5. Subject is a non-smoker for 1 year or greater (if former smoker, less than 10 pack years total smoking history).
6. Subject is able to undergo outpatient (same day) bronchoscopy in the opinion of the investigator or per hospital guidelines.
7. Subject has at least 2 days of asthma symptoms in the last 4 weeks.
8. Subject has an AQLQ score during the baseline period of 6.25 or less.

   * NOTE: Subjects on a dosage regimen of 20mg OCS every other day may be included as this is equivalent to an average daily dosage of 10mg.

Exclusion Criteria:

1. Subject is participating in another clinical trial within 6 weeks of the Baseline Period involving respiratory intervention that could affect the outcome measures of this Study.
2. Over the last 7 days of a 4 week medication stable period, subject requirement for rescue medication use other than for prophylactic use for exercise exceeds an average of:

   1. 8 puffs per day of short-acting bronchodilator, or
   2. 4 puffs per day of long-acting rescue bronchodilator, or
   3. 2 nebulizer treatments per day. At the discretion of the Principal Investigator, subjects considered as unstable on baseline medications may have medications adjusted and re-evaluated after a 4 week medication stabilization period.
3. Subject has a post-bronchodilator FEV1 of less than 65%.
4. Subject has a history of life-threatening asthma, defined by past intubation for asthma, or ICU admission for asthma within the prior 2 years.
5. Subject has 3 or more hospitalizations for exacerbations of asthma in the previous year.
6. Subject has had 4 or more infections of lower respiratory tract (LRTI) requiring antibiotics in the past 12 months.
7. Subject has had 4 or more pulses of systemic corticosteroids (tablets, suspension or injection) for asthma symptoms in the past 12 months.
8. Subject has a known sensitivity to medications required to perform bronchoscopy (such as lidocaine, atropine and benzodiazepines).
9. Subject has other respiratory diseases including emphysema, cystic fibrosis, vocal cord dysfunction, mechanical upper airway obstruction, Churg-Strauss syndrome, and allergic bronchopulmonary aspergillosis (asthma, immediate cutaneous reactivity to A. fumigatus, total serum IgE of >1000ng/mL, elevated specific IgE and IgG to A. fumigatus with or without evidence of central bronchiectasis).
10. Subject has segmental atelectasis, lobar consolidation, significant or unstable pulmonary infiltrate, or pneumothorax, confirmed on x-ray.
11. Subject currently has clinically significant cardiovascular disease, including myocardial infarction, angina, cardiac dysfunction, cardiac dysrhythmia, conduction defect, cardiomyopathy, or stroke.
12. Subject has a known aortic aneurysm.
13. Subject has significant co-morbid illness such as cancer, renal failure, liver disease, or cerebral vascular disease.
14. Subject has uncontrolled hypertension (>200mm Hg systolic or >100mm Hg diastolic pressure).
15. Subject has an implanted electrical stimulation device (e.g., a pacemaker, cardiac defibrillator, or deep nerve or deep brain stimulator).
16. Subject has coagulopathy (INR > 1.5).
17. Subject has any other medical condition that would make them inappropriate for study participation, in the Investigator's opinion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2011-04-07 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Bowman, MD, Study Director — Boston Scientific Corporation
Locations (27):
- United States (23):
  - University of Alabama at Birmingham Lung Health Center, Birmingham, Alabama
  - Yale University Center for Asthma and Airway Disease, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - LSU Health Sciences, New Orleans, Louisiana
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - HealthPartners Specialty Center, Lung and Sleep Health, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - DuBois Regional Medical Center, DuBois, Pennsylvania
  - Pennsylvania State Hershey, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - Franciscan Research Center (St. Joseph Medical Center), Tacoma, Washington
  - MultiCare Pulmonary Specialists, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (4):
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, University of British Columbia, Vancouver, British Columbia
  - Montreal Chest Institute, Montreal, Quebec
  - Hospital Laval Centre de Pneumologie, Sainte-Foy, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Following Last Patient Out, when Results are posted.

REFERENCES:
- [Derived] Chupp G, Kline JN, Khatri SB, McEvoy C, Silvestri GA, Shifren A, Castro M, Bansal S, McClelland M, Dransfield M, Trevor J, Kahlstrom N, Simoff M, Wahidi MM, Lamb CR, Ferguson JS, Haas A, Hogarth DK, Tejedor R, Toth J, Hey J, Majid A, LaCamera P, Fitzgerald JM, Enfield K, Grubb GM, McMullen EA, Olson JL, Laviolette M. Bronchial Thermoplasty in Patients With Severe Asthma at 5 Years: The Post-FDA Approval Clinical Trial Evaluating Bronchial Thermoplasty in Severe Persistent Asthma Study. Chest. 2022 Mar;161(3):614-628. doi: 10.1016/j.chest.2021.10.044. Epub 2021 Nov 10. PMID 34774528
- See also: Bronchial Thermoplasty — http://www.btforasthma.com/

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Procedure
Groups:
- Alair: Participants consented for treatment with Alair
Period: Overall Study
Arm/Group | Alair
Started | 284; 279 Procedure
Completed | 227; 227 Procedure
Not Completed | 57; 52 Procedure
Not completed — Lost to Follow-up | 31
Not completed — Withdrawal by Subject | 14
Not completed — Physician Decision | 8
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Subjects with at least 1 BT procedure.
Arm/Group | Alair
Number analyzed (Participants) | 279
Age, Continuous [Mean (Full Range); unit: years] | 45.71 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 3
  Asian | 4
  Black, of African Heritage | 25
  Caucasian | 234
  Hispanic or Latino | 8
  Other | 5
Height [Mean (Full Range); unit: cm] | 167.4 [133 to 195]
Weight [Mean (Full Range); unit: kg] | 90.3 [49 to 185.5]
BMI [Mean (Full Range); unit: kg/m2] | 32.2 [18.2 to 61.3]
AQLQ [Mean (Standard Deviation); unit: AQLQ Score] — There are 32 questions in the Asthma Quality of Life Questionnaire (AQLQ) and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains.
  AQLQ Score | 4.03 (1.28)
FEV1 - % Predicted [Mean (Standard Deviation); unit: % Predicted]
  Pre-bronchodilator FEV1 | 80.4 (13.7)
  Post-bronchodilator FEV1 | 85.8 (13.6)
Prior 12 months - % Subjects [Count of Participants; unit: Participants]
  Severe Exacerbations | 217
  Hospitalization for asthma | 45
  ER visits for asthma | 82
Prior 12 months - Event rates [Mean (Standard Deviation); unit: # events / subject]
  Severe Exacerbations | 1.61 (1.12)
  Hospitalizations for asthma | 0.22 (0.53)
  ER visits for asthma | 0.54 (1.20)

OUTCOME MEASURES:

1. Primary Outcome: Subjects Experiencing Severe Exacerbations (Rates)
Description: The primary endpoint will be the proportion of subjects experiencing severe exacerbations during the subsequent 12-month (for Years 2, 3, 4, and 5) compared to the first 12-month after the Alair treatment.
Time Frame: Year 1 vs. Year 2, 3, 4, 5
Population: Primary Endpoint - the proportion of subjects experiencing severe exacerbations during the subsequent 12-month (for Years 2, 3, 4, and 5) compared to the first 12-month after the Alair treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Year 1: Proportion of Severe Exacerbations at Year 1
- Year 2: Proportion of Severe Exacerbations at Year 2
- Year 3: Proportion of Severe Exacerbations at Year 3
- Year 4: Proportion of Severe Exacerbations at Year 4
- Year 5: Proportion of Severe Exacerbations at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 262 | 252 | 247 | 240 | 227
Participants | 132 | 118 | 118 | 106 | 97
Statistical Analysis 1: Comparison: Year 1 vs Year 2; Comparison of Years 1 and 2; Test type: Non-Inferiority — An upper 95% confidence limit of the difference between Year 2 compared to the first 12-month proportion is less than 20% will demonstrate that the proportions are not substantially worse during each of the subsequent evaluation periods; Difference of proportions = -0.0380, 95% CI 2-sided [-0.1251 to 0.0497]
Statistical Analysis 2: Comparison: Year 1 vs Year 3; Comparison of Years 1 and 3; Test type: Non-Inferiority — An upper 95% confidence limit of the difference between Year 3 compared to the first 12-month proportion is less than 20% will demonstrate that the proportions are not substantially worse during each of the subsequent evaluation periods; Difference of proportions = -0.0325, 95% CI 2-sided [-0.1197 to 0.0565]
Statistical Analysis 3: Comparison: Year 1 vs Year 4; Comparison of Years 1 and 4; Test type: Non-Inferiority — An upper 95% confidence limit of the difference between Year 4 compared to the first 12-month proportion is less than 20% will demonstrate that the proportions are not substantially worse during each of the subsequent evaluation periods; Difference of proportions = -0.0566, 95% CI 2-sided [-0.1444 to 0.0329]
Statistical Analysis 4: Comparison: Year 1 vs Year 5; Comparison of Years 1 and 5; Test type: Non-Inferiority — An upper 95% confidence limit of the difference between Year 5 compared to the first 12-month proportion is less than 20% will demonstrate that the proportions are not substantially worse during each of the subsequent evaluation periods; Difference of proportions = -0.0765, 95% CI 2-sided [-0.1661 to 0.0130]

2. Secondary Outcome: Rates of Severe Exacerbations
Description: # Severe exacerbations / subject / year
Time Frame: Year 1-5
Measure: Mean (Standard Deviation); unit: # Severe Exacerbations / subject / year
Groups:
- Year 1: Rates of Severe Exacerbations at Year 1
- Year 2: Rates of Severe Exacerbations at Year 2
- Year 3: Rates of Severe Exacerbations at Year 3
- Year 4: Rates of Severe Exacerbations at Year 4
- Year 5: Rates of Severe Exacerbations at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 262 | 252 | 247 | 240 | 227
# Severe Exacerbations / subject / year | 0.93 (1.35) | .92 (1.21) | .77 (1.01) | .84 (1.23) | .72 (1.13)

3. Secondary Outcome: Respiratory Adverse Event Rates
Description: A respiratory adverse event is defined as any sign, symptom, illness, clinically significant abnormal laboratory value, or other adverse medical event associated with the "Respiratory System" that appears or worsens in a subject during a clinical study, regardless of whether or not it is considered related to the procedure used as part of the protocol.
Time Frame: Year 1-5
Measure: Mean (Standard Deviation); unit: # Resp. AE / subject / year
Groups:
- Year 1: Respiratory adverse events at Year 1
- Year 2: Respiratory adverse events at Year 2
- Year 3: Respiratory adverse events at Year 3
- Year 4: Respiratory adverse events at Year 4
- Year 5: Respiratory adverse events at Year
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 276 | 262 | 250 | 240 | 235
# Resp. AE / subject / year | 1.70 (1.95) | 1.52 (1.66) | 1.28 (1.42) | 1.35 (1.63) | 1.22 (1.92)

4. Secondary Outcome: Subjects With Respiratory Adverse Events
Description: as for outcome 3
Time Frame: Year 1-5
Measure: Count of Participants; unit: Participants
Groups:
- Year 5: Respiratory adverse events at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 276 | 262 | 250 | 240 | 235
Participants | 184 | 165 | 155 | 141 | 133

5. Secondary Outcome: Emergency Room Visits for Respiratory Symptoms Rates
Description: Emergency room visits for respiratory symptoms (rates of emergency room visits)
Time Frame: Year 1-5
Measure: Mean (Standard Deviation); unit: # ER Visit / subject / year
Groups:
- Year 1: Emergency room visits for respiratory symptoms rates at Year 1
- Year 2: Emergency room visits for respiratory symptoms rates at Year 2
- Year 3: Emergency room visits for respiratory symptoms rates at Year 3
- Year 4: Emergency room visits for respiratory symptoms rates at Year 4
- Year 5: Emergency room visits for respiratory symptoms rates at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 262 | 252 | 247 | 240 | 227
# ER Visit / subject / year | .31 (.87) | .24 (.80) | .21 (.65) | .17 (.56) | .13 (0.49)

6. Secondary Outcome: Subjects With Emergency Room Visits for Respiratory Symptoms
Description: Subjects with Emergency room visits for respiratory symptoms
Time Frame: Year 1-5
Measure: Count of Participants; unit: Participants
Groups:
- Year 1: Emergency room visits for respiratory symptoms proportions at Year 1
- Year 2: Emergency room visits for respiratory symptoms proportions at Year 2
- Year 3: Emergency room visits for respiratory symptoms proportions at Year 3
- Year 4: Emergency room visits for respiratory symptoms proportions at Year 4
- Year 5: Emergency room visits for respiratory symptoms proportions at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 262 | 252 | 247 | 240 | 227
Participants | 48 | 37 | 32 | 28 | 18

7. Secondary Outcome: Hospitalizations for Respiratory Symptoms Rates
Description: (# hospitalizations for respiratory symptoms / subject / year)
Time Frame: Year 1-5
Measure: Mean (Standard Deviation); unit: # Hospitalizations / subject / year
Groups:
- Year 1: Hospitalizations for respiratory symptoms rates at Year 1
- Year 2: Hospitalizations for respiratory symptoms rates at Year 2
- Year 3: Hospitalizations for respiratory symptoms rates at Year 3
- Year 4: Hospitalizations for respiratory symptoms rates at Year 4
- Year 5: Hospitalizations for respiratory symptoms rates at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 262 | 252 | 247 | 240 | 227
# Hospitalizations / subject / year | 0.13 (0.50) | 0.11 (0.47) | 0.11 (0.47) | 0.05 (0.28) | 0.06 (0.31)

8. Secondary Outcome: Subjects With Hospitalizations for Respiratory Symptoms
Description: Subjects with hospitalizations for respiratory symptoms
Time Frame: Year 1-5
Measure: Count of Participants; unit: Participants
Groups:
- Year 1: Hospitalizations for respiratory symptoms proportions at Year 1
- Year 2: Hospitalizations for respiratory symptoms proportions at Year 2
- Year 3: Hospitalizations for respiratory symptoms proportions at Year 3
- Year 4: Hospitalizations for respiratory symptoms proportions at Year 4
- Year 5: Hospitalizations for respiratory symptoms proportions at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 262 | 252 | 247 | 240 | 227
Participants | 21 | 19 | 18 | 8 | 11

9. Secondary Outcome: Respiratory Serious Adverse Events Rates
Description: The rate of subjects with respiratory serious adverse events (SAEs)
Time Frame: Year 1-5
Measure: Mean (Standard Deviation); unit: # Respiratory SAEs / subect / year
Groups:
- Year 1: Respiratory Serious Adverse Events rates at Year 1
- Year 2: Respiratory Serious Adverse Events rates at Year 2
- Year 3: Respiratory Serious Adverse Events rates at Year 3
- Year 4: Respiratory Serious Adverse Events rates at Year 4
- Year 5: Respiratory Serious Adverse Events rates at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 276 | 262 | 250 | 240 | 235
# Respiratory SAEs / subect / year | 0.14 (0.50) | 0.11 (0.37) | 0.10 (0.41) | 0.06 (0.33) | 0.06 (0.28)

10. Secondary Outcome: Subjects With Respiratory Serious Adverse Events
Description: Subjects with Respiratory Serious Adverse Events
Time Frame: Year 1-5
Measure: Count of Participants; unit: Participants
Groups:
- Year 1: Respiratory Serious Adverse Events proportions at Year 1
- Year 2: Respiratory Serious Adverse Events proportions at Year 2
- Year 3: Respiratory Serious Adverse Events proportions at Year 3
- Year 4: Respiratory Serious Adverse Events proportions at Year 4
- Year 5: Respiratory Serious Adverse Events proportions at Year 5
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 276 | 262 | 250 | 240 | 235
Participants | 26 | 25 | 17 | 10 | 11

11. Secondary Outcome: Pre-bronchodilator FEV1
Description: % Predicted Pre-bronchodilator FEV1
Time Frame: Year 1-5
Measure: Mean (Standard Deviation); unit: % Predicted
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 258 | 235 | 235 | 212 | 217
% Predicted | 89.6 (14.5) | 89.3 (14.6) | 87.7 (14.9) | 88.5 (13.8) | 87.4 (14.6)

12. Secondary Outcome: Post-bronchodilator FEV1
Description: % Predicted Post-bronchodilator FEV1
Time Frame: Year 1-5
Measure: Mean (Standard Deviation); unit: % Predicted
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Number analyzed (Participants) | 257 | 233 | 229 | 212 | 213
% Predicted | 93.1 (13.9) | 92.3 (14.1) | 91.8 (14.2) | 91.1 (14.4) | 91.0 (14.3)

ADVERSE EVENTS:
Time Frame: 5 Years
Description: Adverse events were collected from the time of first BT procedure through the 5-year follow-up.
Arm/Group | Alair
All-Cause Mortality (participants affected / at risk) | 4/279
Serious Adverse Events (participants affected / at risk) | 130/279
Other Adverse Events (participants affected / at risk) | 268/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alair (N=279)
Asthma (Respiratory, thoracic and mediastinal disorders) | 58 (135)
Pneumonia (Infections and infestations) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7)
Influenza (Infections and infestations) | 5 (7)
Bronchitis (Infections and infestations) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Non-cardiac chest pain (General disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Chest pain (General disorders) | 3 (3)
Hiatus hernia (Gastrointestinal disorders) | 3 (3)
Diverticulitis (Infections and infestations) | 3 (3)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (2)
Delivery (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Bipolar I disorder (Psychiatric disorders) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2)
Lung abscess (Infections and infestations) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Tooth malformation (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1)
Excessive skin (Skin and subcutaneous tissue disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Aspergilloma (Infections and infestations) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1)
Caesarean section (Surgical and medical procedures) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alair (N=279)
Asthma (Respiratory, thoracic and mediastinal disorders) | 234 (1258)
Upper respiratory tract infection (Infections and infestations) | 118 (205)
Bronchitis (Infections and infestations) | 89 (152)
Sinusitis (Infections and infestations) | 64 (140)
Cough (Respiratory, thoracic and mediastinal disorders) | 54 (78)
Acute sinusitis (Infections and infestations) | 48 (80)
Oral candidiasis (Infections and infestations) | 40 (71)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 40 (63)
Influenza (Infections and infestations) | 38 (48)
Pneumonia (Infections and infestations) | 37 (49)
Chest pain (General disorders) | 33 (40)
Nasopharyngitis (Infections and infestations) | 28 (42)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (29)
Urinary tract infection (Infections and infestations) | 23 (41)
Headache (Nervous system disorders) | 22 (28)
Lower respiratory tract infection (Infections and infestations) | 19 (26)
Nausea (Gastrointestinal disorders) | 18 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (23)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 17 (21)
Hypertension (Vascular disorders) | 16 (19)
Hypersensitivity (Immune system disorders) | 16 (17)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Chest discomfort (General disorders) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT01350336/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2012-04-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT01350336/Prot_ICF_001.pdf